CLINICAL TRIAL: NCT07034248
Title: Electrochemical Biosensor Based on Lectin-functionalized Nitrogen, Sulfur-doped Graphene Quantum Dot Decorated Gold Nanoparticles for Breast Cancer Diagnosis: From Academic Research to Clinical Translation
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202400729B0
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Electrochemically Sensing Prob; Breast Cancer Diagnosis
Keywords: Electrochemically sensing prob; sulfur-doped graphene quantum dots; breast cancer diagnosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: healthy donors
  Interventions: Other: Electrochemical biosensor
- experimental: breast cancer participants
  Interventions: Other: Electrochemical biosensor

INTERVENTIONS:
Other: Electrochemical biosensor — considering benefits of the nitrogen, sulfur-doped graphene quantum dot (NSGQDs) and 3-dimensional gold nanoparticle (AuNP), we used these materials for the construction of a novel electrochemical biosensor to apply the synergy contributions on the enhancement of the potential in clinical and cancer diagnostic applications. The synthesis of a novel nanocomposite through the integration of NSGQDs with AuNP yields a hybrid material (NSGQDs/AuNP) that combines the advantages of both its organic and inorganic properties, potentially revealing unique characteristics to enhance the electrochemical behaviors, which establishes a robust foundation for constructing a label-free electrochemical biosensor. This pioneering biosensor was then conjugated with PhaL (NSGQDs/AuNP/PhaL) through the amide bond between the COOH group of NSGQDs and the NH2 group of PhaL, which has the potential for the ultra-sensitive detection of cancer markers, featuring heightened electrochemical and sensing capabilitie

SUMMARY:
In this research, considering benefits of the nitrogen, sulfur-doped graphene quantum dot (NSGQDs) and 3-dimensional gold nanoparticle (AuNP), we used these materials for the construction of a novel electrochemical biosensor to apply the synergy contributions on the enhancement of the potential in clinical and cancer diagnostic applications. The synthesis of a novel nanocomposite through the integration of NSGQDs with AuNP yields a hybrid material (NSGQDs/AuNP) that combines the advantages of both its organic and inorganic properties, potentially revealing unique characteristics to enhance the electrochemical behaviors, which establishes a robust foundation for constructing a label-free electrochemical biosensor. This pioneering biosensor was then conjugated with PhaL (NSGQDs/AuNP/PhaL) through the amide bond between the COOH group of NSGQDs and the NH2 group of PhaL, which has the potential for the ultra-sensitive detection of cancer markers, featuring heightened electrochemical and sensing capabilities that make substantial contributions to the field of cancer detection. The detection principle of breast cancer is based on the change in impedance of NSGQDs/AuNP/PhaL after the addition of breast cancer cell, which can inhibit the electron transfer after the formation of breast cancer cell bioconjugate with NSGQDs/AuNP/PhaL. NSGQDs/AuNP/PhaL are used as the bi-functional probe to amplify the electrochemical activity as well as to link cancer cell. The developed novel NSGQDs/AuNP/PhaL biosensor show high sensitivity and good stability for quantitative determination of breast cancer cell in a linear range of 5 - 2500 cell mL-1 with limit of detection (LOD) of 6 cancer cell mL-1, which exhibits a great potential in clinical and cancer diagnostic applications. The superior sensitivity of the developed impedimetric immunosensor is mainly attributed to the remarkable electro-conductivity of NSGQDs/AuNP, which can accelerate the electron transfer process between NSGQDs/AuNP/PhaL and electrolyte. This achievement paves the way for the development of a lectin-based sensing probe as a robust platform for the ultrasensitive and selective detection of MCF-7 and other cancer cell lines. Such advancements hold significant promise for facilitating early diagnosis and therapy of diseases, particularly in the context of breast cancer.

DETAILED DESCRIPTION:
Breast cancer can develop when cells in the breast tissue undergo uncontrollable growth due to genetic, hormonal, environmental, and lifestyle factors. Genetic mutations, particularly in genes like BRCA1 and BRCA2, can increase susceptibility to breast cancer. In addition, hormonal influences, such as prolonged exposure to estrogen and progesterone, also contribute to cell proliferation. Environmental exposures, like radiation, along with lifestyle factors such as obesity and alcohol consumption, further elevate the risk. Abnormalities in cell growth and DNA damage can lead to the formation of tumors within the breast tissue. While some tumors may be benign, others can be malignant and potentially spread to other parts of the body [6]. It is important to note that not all breast tumors or abnormalities lead to cancer, and many breast cancers are treatable, especially when detected early through screening.

The rising complexity of diagnosing and treating breast cancer poses challenges across all resource settings. The advancement of cancer diagnosis systems is an urgent task for Worldwilde Health Organiation [7]. Implementing population-based screening programs for the early detection of asymptomatic disease emerges as a sensible strategy to reduce mortality. Nevertheless, these initiatives are costly and demand substantial resources. They also necessitate the establishment of comprehensive and quality-assured cancer services to effectively treat the identified diseases.

1.3. Conventional methods for breast cancer detection The traditional approach to breast cancer detection typically involves a combination of clinical breast examinations, imaging, and biopsy procedures. These methods have been the cornerstone of breast cancer screening for decades and have proven effective in detecting abnormalities in breast tissue [8, 9]. One of the most popular breast cancer detection methods is mammography. Mammograms are X-ray images of the breast that can detect early signs of breast cancer, such as lumps or calcifications, before they can be felt through a breast exam. Mammography is recommended as a screening tool for women starting at age 40, and it is considered the gold standard for detecting breast cancer in its early stages. Additionally, ultrasound and magnetic resonance imaging (MRI) may be used in conjunction with mammography for further evaluation or screening in certain cases, especially for women at higher risk or with dense breast tissue. Other popular methods include clinical breast examinations (CBE), where a healthcare provider manually examines the breasts for abnormalities, and breast self-exams (BSE), where women check their own breasts regularly for any changes. If suspicious abnormalities are detected through clinical examinations or imaging, a biopsy is performed to obtain tissue samples for analysis. There are various biopsy techniques, including: fine-needle aspiration (FNA), core needle biopsy (CNB), and surgical biopsy.

Conventional methods for breast cancer detection have several advantages, such as their proven effectiveness, widespread availability, and the ability to detect cancer at an early stage. They provide clear visualizations of tumors and facilitate tissue diagnosis through procedures like biopsies. Some methods are minimally invasive, reducing patient discomfort. However, these methods have limitations, including the potential for false results, exposure to radiation in imaging techniques, and invasive procedures that carry risks. Certain cancers may not be as effectively detected by these methods, and they can be expensive. Routine screening can lead to overutilization, unnecessary procedures, and patient anxiety. Moreover, these methods lack the precision of molecular information that is increasingly crucial for personalized treatment. They may not be suitable for large-scale population screening, and some cancers may have already metastasized before detection. To address these limitations, ongoing research explores the integration of molecular and genetic data to enhance diagnostic accuracy and tailor treatment decisions to individual patients.

1.4. ELISA for breast cancer detection Enzyme-Linked Immunosorbent Assay (ELISA) is a valuable tool in cancer detection and diagnosis. This highly sensitive and specific laboratory technique is based on the principles of antigen-antibody interaction and can be applied to various cancer-related biomarkers. Principally, ELISA relies on the specific binding of an antigen (a cancer-related protein or biomarker) in a patient's sample to an immobilized antibody on a solid surface. This interaction is then visualized using an enzyme-linked secondary antibody and a substrate that produces a detectable signal. ELISA can be customized to detect specific cancer biomarkers, such as prostate-specific antigen (PSA) for prostate cancer, carcinoembryonic antigen (CEA) for colorectal cancer, or CA-125 for ovarian cancer, and CA15-3 for breast cancer [10, 11]. Elevated levels of these biomarkers in a patient's blood or tissue can indicate the presence of cancer.

ELISA is also known for its high sensitivity, allowing for the detection of cancer at an early stage when treatment is often more effective. Regular monitoring of biomarker levels through ELISA can help in disease surveillance and early intervention, and characterizing tumors by assessing the expression of specific biomarkers associated with different types of cancer. ELISA is a cost-effective, high-throughput method that is widely used in clinical laboratories. Nevertheless, it is not without challenges, as cross-reactivity can result in false results. Thus, rigorous quality control and validation procedures are imperative. In summary, ELISA is an indispensable tool in the diagnosis, early intervention, and ongoing management of cancer, offering a valuable means to identify and monitor the disease and improve patient outcomes.

1.5. Flow cytometry for breast cancer detection Flow cytometry is a versatile and robust technique with wide applications in cancer detection. It operates by passing cells through a laser-based instrument, enabling the analysis of individual cells based on their physical and chemical properties [12]. In the context of cancer, flow cytometry is particularly useful for identifying cancer cells through the detection of specific cell surface markers. Antibodies labeled with fluorescent dyes bind to these markers, allowing for precise quantification [13]. Moreover, flow cytometry aids in subtyping and characterizing cancer types by evaluating the expression of particular proteins, which is a crucial step in personalized treatment decisions.

Flow cytometry goes beyond surface markers; it can also analyze DNA content within cancer cells, which is vital for identifying aneuploidy, a common characteristic in many cancer types. This technique is exceptionally sensitive, enabling the early detection of cancer cells, even when they are present in low quantities. Flow cytometry is essential for assessing cell viability and apoptosis, providing critical information about how cancer cells are responding to treatment [14]. It is also instrumental in minimal residual disease (MRD) detection, which involves identifying and quantifying remaining cancer cells post-treatment to evaluate the success of therapy and potential relapse risks.

Despite its advantages, including high-throughput capabilities and detailed single-cell analysis, flow cytometry requires skilled operators and specialized instrumentation. Additionally, its effectiveness may depend on the availability of specific antibodies and markers for less common cancer types. Flow cytometry is an invaluable tool in the field of cancer detection, providing precise insights into cancer cell characteristics, subtypes, and viability, thus contributing significantly to both clinical diagnostics and cancer research.

1.6. Electrochemical biosensors for cancer detection Biosensors have emerged as innovative and promising tools for cancer detection. These devices integrate biological components with transducers to detect specific cancer-related biomarkers or changes in the biological environment. Their ability to detect cancer-specific biomarkers and facilitate real-time tracking makes them valuable tools for early diagnosis, treatment assessment, and personalized cancer care. As technology continues to advance, biosensors are likely to play an increasingly important role in improving cancer outcomes. Biosensors operate on the principle of recognizing and measuring specific biomolecules or biological changes . They often use bioreceptors (e.g., antibodies, enzymes, DNA) that interact with cancer-related molecules.

Optical and electrochemical techniques have been at the forefront of cancer detection, offering high sensitivity. Especially, electrochemical sensors have emerged as powerful tools in the realm of cancer detection, offering innovative and highly sensitive approaches for the identification and quantification of cancer-related biomarkers [15]. These sensors harness the principles of electrochemistry to convert biochemical interactions at the sensor surface into measurable electrical signals, making them valuable assets in the early diagnosis and monitoring of cancer. Electrochemical sensors provide a means to detect and analyze the specific biomolecules or biomarkers in the body with remarkable sensitivity and specificity. Electrochemical biosensors have demonstrated potential for detecting a wide range of cancer biomarkers, including proteins, nucleic acids, and tumor-specific metabolites, offering non-invasive or minimally invasive approaches for early cancer diagnosis, monitoring treatment response, and detecting cancer recurrence (Fig. 2). Examples of specific cancer-related applications include the detection of prostate-specific antigen (PSA) for prostate cancer, carcinoembryonic antigen (CEA) for colorectal cancer, CA15-3 for breast cancer and various genetic mutations associated with different cancer types [16, 17].

Fig. 2. Electrochemical sensors for the early diagnosis of diverse breast cancer biomarkers [17].

Various electrochemical techniques, including voltammetry, impedance spectroscopy, and electrochemical impedance spectroscopy, are utilized for signal transduction. The most classical application of electrochemical biosensors in the early diagnosis of tumors is the detection of tumor cells by biosensors based on cell impedance sensing technology [15]. In addition, cyclic voltammetry (CV), as a commonly used electrochemical research method, can be used to judge the microscopic reaction process on the electrode surface, so as to detect the change in impedance or microcurrent at the electrode interface caused by the growth of cells on the electrode surface. Differential pulse voltammetry (DPV) is a method based on linear sweep voltammetry (LSV) and staircase voltammetry which has a lower background current and higher detection sensitivity. In addition, it displays the highly stable and specific capture of cancer cells by producing nontoxic biological modifications on the working electrodes of electrochemical biosensors, such as with covalently linked biotin, monoclonal antibodies, lactoglobulin A and aptamer. Therefore, the detection of tumor cells without lysis and fixation is made possible, which simplifies the analysis process and improves the accuracy of the results. Ongoing research aims to further optimize the sensitivity, specificity, and reliability of electrochemical biosensors for robust and cost-effective cancer detection in clinical settings [18, 19].

1.6.1. Electrode material The choice of electrode material is a crucial aspect in the design and performance of electrochemical biosensors. Electrodes play a fundamental role in facilitating electron transfer during electrochemical reactions, and the selection of an appropriate material directly impacts the sensitivity, stability, and overall efficiency of the electrochemical biosensor. Several materials are commonly used as electrode materials in electrochemical biosensors, each with its unique properties and advantages. The choice of electrode material depends on the specific application and the nature of the analyte being detected (Table 1). The Au, Pt, Ag electrodes are extensively employed as electrode materials due to their excellent conductivity, chemical stability, and biocompatibility [20]. These nanomaterials surfaces are not only easily modified with self-assembled monolayers (SAMs) but also immobilize biomolecules effectively. Additionally, gold nanoparticles (AuNP) are also popular for enhancing the surface area and improving the electrocatalytic activity.

Nevertheless, carbon-based materials are widely utilized as electrode materials in electrochemical biosensors due to their exceptional properties, including high electrical conductivity, large surface area, and biocompatibility [21]. Graphene, a single layer of carbon atoms arranged in a hexagonal lattice, stands out for its high surface area, exceptional electrical conductivity, and biocompatibility, making it an ideal platform for efficient electron transfer and biomolecule immobilization [22]. Carbon nanotubes, cylindrical structures of rolled-up graphene sheets, provide high conductivity and a large surface area, enhancing biosensor performance. Carbon nanofibers, with their high electrical conductivity and stability, contribute to improved biosensor sensitivity and selectivity. Glassy carbon, known for its amorphous structure, offers good electrical conductivity and chemical stability, making it widely used in various biosensing applications. Additionally, activated carbon, a porous material with a large surface area, is often combined with other electrode materials to enhance biomolecule adsorption and improve biosensor sensitivity. The choice of carbon electrode material depends on specific biosensing requirements, allowing researchers to tailor these materials for applications ranging from medical diagnostics to environmental monitoring [23].

Graphene quantum dots (GQDs), also known as semiconductor nanocrystal, has been a hot new type of luminescent carbon-based nanomaterials in recent years, with unique optical and electrical properties, which stand out as promising electrode materials for electrochemical biosensors. Derived from graphene, GQDs offer a high surface area, excellent electrical conductivity, and biocompatibility, enhancing biosensor sensitivity [24]. Their quantum confinement effects result in size-dependent optical and electronic properties, advantageous for fluorescence-based biosensing. GQDs' tailorable surface chemistry allows for specific biomolecule binding, ensuring selective target detection. With low toxicity and potential photoluminescence properties, GQDs provide a versatile platform for constructing biosensors with applications in medical diagnostics, environmental monitoring, and food safety [25]. Researchers are actively exploring and optimizing the use of GQDs to advance biosensor performance. While GQDs inherently exhibit semiconductor properties, their remarkable electrical characteristics, particularly the high electron mobility and ballistic transport of charge carriers facilitated by the sp2-hybridized two-dimensional single-atom thick-layer structure, render them exceptionally appealing for electrochemical sensing applications. The incorporation of metal nanoparticles into GQDs has recently garnered considerable attention in research. This interest is driven by the emergence of novel and/or enhanced functionalities that result from the synergistic combination of these components, which holds significant promise for diverse applications, including electro-catalysis and optoelectronic capabilities. Furthermore, the introduction of heteroatoms such as N, S, and B into GQDs can significantly augment the electron density on the surface framework, thereby enhancing sensing sensitivity and selectivity for a wide range of analyte detections. The synthesis of a novel nanocomposite by combining NSGQDs with AuNP results in a hybrid material that combines the advantages of both organic and inorganic components, potentially showcasing unique properties. Moreover, incorporating NSGQDs onto AuNP nanocomposites provides a compelling platform for the development of a label-free electrochemical biosensor, which holds the potential for ultra-sensitive detection of cancer markers, offering enhanced electrochemical and sensing capabilities that contribute significantly to the field of cancer detection.

Table 1. Performance metrics of previously documented electrochemical biosensors for detecting breast cancer biomarkers.

Analyte Detection technique Nanomaterials Performance Ref. MCF-7 Electrochemical impedance (EIS) Au nanoparticles (AuNPs) LOD: 10 cells/mL [26]

Hela Electrochemical impedance (EIS) Multiwall carbon nanotubes (MWCNTs) Linear range: 2.1 x 102-2.1 x 107 cells/mL LOD: 70 cells/mL [27]

HL-60 Cyclic voltammetry (CV) Electrochemical impedance (EIS) Differential pulse voltammetry (DPV) Multiwall carbon nanotubes (MWCNTs) Linear range: 2.7 x 102-2.7 x 107 cells/mL LOD: 90 cells/mL [28]

K562 Cyclic voltammetry (CV) Electrochemical immunosensors Au nanoparticles (AuNPs) Linear range: 1.0 x 102-1.0 x 107 cells/mL [29]

MCF-7 Electrochemical nucleic acid biosensors DNA-AgNC LOD: 3 cells/mL [30]

MCF-7 Electrochemical nucleic acid biosensors Multi-wall carbon nanotubes (MWCNTs) Linear range: 1.0 x 102-1.0 x 107 cells/mL LOD: 25 cells/mL [31]

CTCs Cyclic voltammetry (CV) Electrochemical impedance (EIS) Pt@Ag nanoflower AuNPs/Acetylene black Linear range: 20-106 cells/mL LOD: 3 cells/mL [32]

CTCs Cyclic voltammetry (CV) Differential pulse voltammetry (DPV) Electrochemical impedance Magnetic Fe3O4 nanospheres (MNs) Cu2O nanoparticles (Cu2O NPs) Linear range: 3.0-3000 cells/mL LOD: 1 cells/mL [33]

CTCs (MCF-7) Cyclic voltammetry (CV) Electrochemical impedance (EIS) Ni micropillars/ PLGA electrospun Nanofibers Linear range: 10-105 cells/mL LOD: 8 cells/mL [34]

K562 Differential pulse voltammetry (DPV) Graphene oxide/ quantum dots (QDs) LOD: 60 cells/mL [35]

HepG2 Electrochemical impedance (EIS) Carbon nanotubes (CNTs) Linear range: 10-105 cells/mL [36]

CTCs Cyclic voltammetry (CV) Electrochemical impedance (EIS) Au-wire Linear range: 30-106 cells/mL LOD: 10 cells/mL [37]

HT 29 FR-positive cancer cells Electrochemical Functionalized fibrous Nanosilica (KCC-1) Linear range: 50-1 x 1.2 x 104 cells/mL LOD: 50 cells/mL [7]

1.6.2. Cyclic voltametry (CV) in electrochemical biosensor Cyclic voltammetry (CV) is a fundamental electrochemical technique widely employed in the development and characterization of electrochemical biosensors. Within the realm of biosensors, which integrate a biological recognition element with a transducer for converting biological responses into measurable electrical signals, CV assumes a pivotal role. In the CV process, a potential waveform is systematically applied to an electrochemical cell, and the ensuing current is measured, resulting in a cyclic voltammogram. This voltammogram graphically represents the current response against the applied potential and is particularly insightful for studying the electrochemical behavior of redox-active species. In the context of electrochemical biosensors, where a biorecognition element is immobilized on an electrode surface, CV facilitates the examination of reaction kinetics, thermodynamics, and the optimization of conditions for effective immobilization [38]. Additionally, CV aids in enhancing the sensitivity of biosensors by optimizing signal amplification, while also providing a means to evaluate stability and reproducibility over multiple cycles. The technique serves as a valuable tool for researchers in understanding and refining the electrochemical parameters essential for the reliable detection and quantification of biological analytes in biosensor applications.

1.6.3. Electrochemical impedance spectroscopy (EIS) in electrochemical biosensor Electrochemical impedance spectroscopy (EIS) is a powerful analytical technique employed in the development and characterization of electrochemical biosensors. In contrast to traditional electrochemical methods like CV, EIS provides insights into both the capacitive and resistive characterization of a system over a range of frequencies [17]. This versatility makes EIS particularly valuable for studying the interactions at the electrode-bio-interface in biosensor applications.

EIS involves the application of a small amplitude alternating current (AC) signal to the working electrode, and the resulting impedance response is analyzed across a range of frequencies. The impedance spectrum obtained typically includes information about charge transfer resistance, double-layer capacitance, and solution resistance, offering a more comprehensive understanding of the electrochemical processes occurring at the electrode surface.

1.6.4. Differential pulse voltammetry in electrochemical biosensor Differential pulse voltammetry (DPV) is a technique employed in electrochemical biosensors for the selective detection and analysis of various analytes. This method involves applying a potential pulse to the working electrode while measuring the resulting current. The key feature of DPV is the subtraction of a pre-pulse baseline current from the current measured after the potential pulse, allowing for enhanced sensitivity and selectivity in detecting electroactive species. In the context of electrochemical biosensors, DPV offers distinct advantages [39]. The differential nature of the measurement minimizes background interference, leading to improved signal-to-noise ratios. This makes DPV particularly valuable for the detection of specific biomolecules or analytes in complex biological samples.

The working principle involves scanning the potential at the working electrode, applying a series of voltage pulses, and measuring the resulting current. The current response is then analyzed differentially to enhance the detection of target analytes. DPV is widely utilized in biosensing applications due to its ability to provide quantitative and precise measurements, especially in the presence of interfering substances. The application of DPV in electrochemical biosensors contributes to the broader field of analytical chemistry, offering a versatile and effective tool for the sensitive detection of biomolecules and analytes in various domains, ranging from clinical diagnostics to environmental monitoring.

1.7. Highlight of research In this research, considering benefits of the NSGQDs and AuNP, we used these materials for the construction of a novel electrochemical biosensor to apply the synergy contributions on the enhancement of the potential in clinical and cancer diagnostic applications. The synthesis of a novel nanocomposite through the integration of NSGQDs with AuNP yields a hybrid material that combines the advantages of both its organic and inorganic properties, potentially revealing unique characteristics to enhance the electrochemical behaviors, which establishes a robust foundation for constructing a label-free electrochemical biosensor. This pioneering biosensor has the potential for the ultra-sensitive detection of cancer markers, featuring heightened electrochemical and sensing capabilities that make substantial contributions to the field of cancer detection.

The detection principle of breast cancer is based on the change in impedance of NSGQDs@AuNP after the addition of breast cancer cell, which can inhibit the electron transfer after the formation of breast cancer cell bioconjugate on the NSGQDs/AuNP surface. As shown in Fig. 4 NSGQDs and NSGQDs/AuNP are fabricated by the hydrothermal pyrolysis and reduction methods, respectively. NSGQDs/AuNP are used as the bi-functional probe to amplify the electrochemical activity as well as to link cancer cell. The developed novel NSGQDs@AuNP nanocomposites show high sensitivity and good stability for quantitative determination of breast cancer cell in a linear range of 5 - 2500 cell mL-1 with limit of detection (LOD) of 6 cell mL-1, which exhibits a great potential in clinical and cancer diagnostic applications. The superior sensitivity of the developed impedimetric immunosensor is mainly attributed to the remarkable electro-conductivity of NSGQDs@AuNP, which can accelerate the electron transfer process between NSGQDs and electrode.

ELIGIBILITY:
Inclusion Criteria:

* age 18-90
* health participants: without cancer over 5 years
* cancer participants: diagnosis of breast cancer
* cancer participants: agree to receive treatment in Chang Gung hospital

Exclusion Criteria:

* mental disease
* Physician's assessment not suitable

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in two branch hospitals of Chang Gung Memorial Hospital, Taiwan including Linkou and Tucheng. Healthy and breast cancer participants.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity and selectivity on electrochemical biosensor | From enrollment to the following 3 years
  The detection principle of breast cancer is based on the change in impedance of NSGQDs@AuNP after the addition of breast cancer cell, which can inhibit the electron transfer after the formation of breast cancer cell bioconjugate on the NSGQDs/AuNP surface.
  NSGQDs and NSGQDs/AuNP are fabricated by the hydrothermal pyrolysis and reduction methods, respectively. NSGQDs/AuNP are used as the bi-functional probe to amplify the electrochemical activity as well as to link cancer cell. The developed novel NSGQDs@AuNP nanocomposites show high sensitivity and good stability for quantitative determination of breast cancer cell in a linear range of 5 - 2500 cell mL-1 with limit of detection (LOD) of 6 cell mL-1

CONTACTS AND LOCATIONS:
Overall Officials: CHIA-HSUN Hsieh, M.D PhD, Principal Investigator — Chang Gung Memorial Hospital